CLINICAL TRIAL: NCT04357015
Title: Comparative Safety and Efficacy of Intravenous Tranexamic Acid Versus IV Carbetocin in Reducing Blood Loss During Abdominal Myomectomy: a Randomized Controlled Trial
Brief Title: Intravenous Tranexamic Acid Versus IV Carbetocin in Abdominal Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: tranexamic acid myomectomy
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Myomectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intravenous tranexamic acid (Experimental): The tranexamic acid (TXA) group will receive a single bolus IV injection of 15 mg/kg of TXA 20 minutes before surgical incision
  Interventions: Drug: intravenous tranexamic acid
- intravenous carbetocin (Active Comparator): The carbetocin group will receive a single bolus IV injection of 100 mcg of carbetocin 20 minutes before surgical incision
  Interventions: Drug: intravenous carbetocin
- placebo (Placebo Comparator): the placebo group will be given a normal saline IV bolus 20 minutes before surgical incision
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: intravenous tranexamic acid — The tranexamic acid (TXA) group will receive a single bolus IV injection of 15 mg/kg of TXA 20 minutes before surgical incision
  Arms: intravenous tranexamic acid
Drug: intravenous carbetocin — The carbetocin group will receive a single bolus IV injection of 100 mcg of carbetocin 20 minutes before surgical incision
  Arms: intravenous carbetocin
Drug: placebo — the placebo group will be given a normal saline IV bolus 20 minutes before surgical incision
  Arms: placebo

SUMMARY:
the aim of the present study is to compare safety and efficacy of intravenous tranexamic acid versus IV carbetocin in reducing blood loss during abdominal myomectomy: a randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* women with symptomatic fibroids candidate for abdominal myomectomy with staging of myoma from (3 to 6) according to FIGO staging

Exclusion Criteria:

* women with Myoma FIGO staging (1,2,7 and 8) candidate for laparoscopic or hysteroscopic myomectomy, women with allergy or contraindications to carbetocin or tranexamic acid

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-10-10 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | one hour
  the intraoperative blood loss in ml will be estimated during the procedure

SECONDARY OUTCOMES:
need for blood transfusion | 24 hours
  need for intraoperative or postoperative blood transfusion